CLINICAL TRIAL: NCT02922257
Title: Prospective, Non-interventional Clinical Study of Biomarker Expression in Patients With ACTH-Dependent Cushing's Syndrome Before and After Surgery
Brief Title: Biomarker Expression in Patients With ACTH-Dependent Cushing's Syndrome Before and After Surgery
Status: Completed | Type: Observational
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: FKBP5-700
Record Dates: First submitted 2016-09-27; First posted 2016-10-04 (Estimated); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Cushing's Syndrome
MeSH Terms: conditions — Cushing Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — RNA extracted from blood samples
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will investigate the potential for FK506 binding protein 5 (FKBP5) (and other gene expression markers, for example pentraxin 3 [PTX-3], serum/glucocorticoid regulated kinase 1 [SGK1], and glycogen synthase kinase 3 beta [GSK3b]) to be developed as a biomarker for use in diagnosis of Cushing's syndrome, assessment of effectiveness of medical or surgical treatment, and detection of relapse of endogenous Cushing's syndrome after surgery.

DETAILED DESCRIPTION:
This study will investigate the potential for FK506 binding protein 5 (FKBP5) (and other gene expression markers, for example pentraxin 3 [PTX-3], serum/glucocorticoid regulated kinase 1 [SGK1], and glycogen synthase kinase 3 beta [GSK3b]) to be developed as a biomarker for use in diagnosis of Cushing's syndrome, assessment of effectiveness of medical or surgical treatment, and detection of relapse of endogenous Cushing's syndrome after surgery.

The primary study hypothesis is that FKBP5 levels are elevated in patients with Cushing's syndrome, and these levels decrease after successful surgical treatment.

This is a non-randomized specimen collection study with pre- and post-surgery follow-up periods. This study will be performed in patients with adrenocorticotropic hormone (ACTH)-dependent Cushing's syndrome scheduled for curative surgery and followed until relapse of endogenous Cushing's syndrome or up to 3 years post-surgery. No study medication will be given.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age.
* Has a documented diagnosis of ACTH-dependent, endogenous Cushing's syndrome and is scheduled for curative surgery.
* Must be able to comprehend and sign an approved Informed Consent Form (ICF) and other applicable study enrollment documents.

Exclusion Criteria:

* Plans for pre-operative and/or intra-operative use of glucocorticoid ("steroid cover").
* Use any of the following treatments for Cushing's syndrome, as specified:
* 4 weeks prior to first specimen collection and/or during the study period.

  * Adrenostatic medications (metyrapone, ketoconazole, fluconazole, aminoglutethimide, LCI699 or etomidate etc).
  * Short-acting somatostatin analogs (octreotide, pasireotide).
* 6 weeks prior to first specimen collection and/or during the study period.

  o Mifepristone.
* 8 weeks prior to first specimen collection and/or during the study period.

  o Neuromodulator drugs that act at the hypothalamic-pituitary level: serotonin antagonists (cyproheptadine, ketanserin, retanserin), dopamine agonists (bromocriptine, cabergoline), gamma-aminobutyric acid agonists (sodium valproate), and somatostatin receptor ligands (octreotide long-acting release [LAR], pasireotide LAR, lanreotide).
* Concomitant use of the following due to their potential to stimulate the expression of FKBP5:
* Testosterone or other steroid hormone analogues.
* Oral contraceptives or hormonal replacement therapy.
* History of illness that the Principal Investigator (PI) considers could interfere with or affect the conduct, results, and/or completion of the clinical trial.
* Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * ≥ 18 years of age both male and female.
  * Has a documented diagnosis of ACTH-dependent, endogenous Cushing's syndrome and is scheduled for curative surgery.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Gene expression levels | three years
  Change in FKBP5 expression levels from baseline to after surgical treatment but prior to glucocorticoid replacement therapy

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Moraitis, M.D., Study Director — Corcept Therapeutics
Locations (4):
- United States (4):
  - Los Angeles, California
  - Rochester, Minnesota
  - Cleveland, Ohio
  - Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided